CLINICAL TRIAL: NCT03924297
Title: Chilipad for Sleep and Symptoms of PTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: eIRB withdrew study for concerns
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00057589
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-04

CONDITIONS: PTSD
Keywords: chilipad
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Twenty subjects with PTSD will use the Chilipad nightly for 5 weeks. The subjects will be given an OURA ring to measure sleep duration and quality during the 5 weeks. Subjects will also be given questionnaires before and after the sleep study part of the study to measure changes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Chilipad Arm (Experimental): Subjects will use chilipad nightly for 5 weeks
  Interventions: Device: chilipad

INTERVENTIONS:
Device: chilipad — Chilipad is a commercially available pad designed to be placed between the top of a mattress and bed sheets. It allows for precise temperature regulation in one's bed.

SUMMARY:
The purpose of this study is to obtain pilot data in preparation for future research designed to formally evaluate the effectiveness of the Chilipad for patients with PTSD

DETAILED DESCRIPTION:
This is a prospective cohort, before-after trial. 20 subjects with PTSD or PTSD symptoms (per patient report) will use the Chilipad nightly for 5 weeks after completing a short battery of PROMIS questionnaires. During the 5-week study intervention, subjects will also wear an OURA ring on a finger. The OURA week measures sleep duration and quality. 5 weeks after study enrollment, patients will repeat the battery or PROMIS questionnaires and will return the Chilipad and OURA rings, both of which will be provided free of charge by the Chilipad and OURA manufacturers

ELIGIBILITY:
Inclusion Criteria:

* Patients who have seen the study PI (Remy Coeytaux, MD, PhD) for an integrative medicine consultation between September 1, 2018 and April 30, 2019 and who report having been diagnoses with PTSD or who believe they may have PTSD or PTSD-related symptoms are eligible to participate.

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
PROMIS Sleep Related Impairment Short Form | 5-week prior intervention
  PROMIS sleep related impairment short form is a questionnaire that ranges in score from 8-40; the lower the score, the better the outcome.
PROMIS Sleep Related Impairment Short Form | 5-week after intervention
  PROMIS sleep related impairment short form is a questionnaire that ranges in score from 8-40; the lower the score, the better the outcome.

SECONDARY OUTCOMES:
PROMIS anxiety short form | 5-week prior intervention
  PROMIS anxiety short form is a questionnaire that ranges in score from 8-40; the lower the score, the better the outcome.
PROMIS Anger Short form | 5-week after intervention
  the PROMIS anger short form is a questionnaire that ranges in score from 5-25; the lower the score, the better the outcome.
OURA ring total sleep metric | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The total sleep metric will show hours of sleep each night.
OURA ring REM metric | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The total REM metric will show the total amount of REM sleep each night.
OURA ring DEEP sleep metric | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The DEEP sleep metric will show the number of hours of deep sleep each night.
OURA ring Efficiency metric | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. Efficiency means the percentage of time spent sleeping while in bed.
OURA ring latency metric | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. Latency is the amount of time it takes a study participant to fall to sleep.
OURA ring timing metric | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The timing records individual circadian rhythms.
OURA ring sleep score metric | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The sleep score metric will be determined by total sleep, efficiency, disturbances, REM sleep, deep sleep, sleep latency, sleep timing and light sleep.The sleep score ranges from 0-100. Higher scores denotes better outcomes.
OURA ring resting heart rate | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The resting heart rate will be recorded.
OURA ring heart rate variability | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The heart rate variability will be recorded.
OURA ring respiration rate | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The respiration rate will be recorded.
OURA ring lowest resting heart rate | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The lowest resting heart rate will be recorded.
OURA ring readiness score | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The readiness score is calculated taking in account sleep balance, previous day activity, activity balance, body temperature, resting heart rate (rhr), recovery index . Score will be between 0 and 100. A lower score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Remy Coeytaux, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: describes oura ring outcome measures in detail — https://ouraring.com/